CLINICAL TRIAL: NCT06385652
Title: Clinical PET Imaging Evaluation of 68Ga-NB381 Probe in Multiple Myeloma
Brief Title: PET Imaging Study of 68Ga-NB381 in Multiple Myeloma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUFH-MM-NB381
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: In this sequential assignment clinical trial, we aim to evaluate and compare the diagnostic performance of two PET imaging agents, 68Ga-NB381 and 18F-FDG, in patients diagnosed with multiple myeloma (MM). The study will enroll MM patients who meet the inclusion criteria and are scheduled for routine diagnostic imaging.
  Each participant will undergo PET imaging with 18F-FDG first, followed by a second PET scan using 68Ga-NB381 (or reversed). To minimize potential interference between the two imaging sessions and ensure patient safety, a minimum interval of one day will be maintained between the two scans, with all imaging completed within one week. This sequential imaging approach allows for direct comparison of the imaging agents in the same patient, thus controlling for inter-patient variability and providing a more accurate assessment of the relative merits of each imaging agent in the same metabolic and pathological condition.
Masking Description: All PET/CT images are jointly interpreted by at least two imaging and nuclear medicine physicians, each with several years of diagnostic experience and at least at the attending physician level. They compare and record the number of lesions detected and the SUVs (Standard Uptake Values) for both 18F-FDG and 68Ga-NB381 PET/CT scans. After consultation, they provide a unified diagnostic opinion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Head to head PET imaging comparison between 18F-FDG and 68Ga-NB381 for MM diagnosis (Experimental): 1. 68Ga-NB381 PET/CT Examination: The patient will be intravenously injected with prepared and quality-controlled 68Ga-NB381 (0.05-0.1 mCi/kg). Two hours post-injection, a full-body scan will be conducted using the Shanghai United Imaging uMI 780 PET/CT, covering from the top of the head to the mid-thigh. If indeterminate lesions are identified in routine imaging, delayed imaging will be performed for further evaluation. The patient should lie in a supine position and breathe calmly. Data will be reconstructed using the OSEM method to obtain coronal, sagittal, and transverse PET and PET/CT fused images.
  2. 18F-FDG PET/CT Examination: Patients must fast for more than 6 hours before the examination. 18F-FDG (0.05-0.1 mCi/kg) will be administered intravenously, and one hour later. Same requirement as mentioned above.
  Interventions: Drug: 68Ga-NB381

INTERVENTIONS:
Drug: 68Ga-NB381 — Lei Kang from Peking University First Hospital and Bing Jia's team from the School of Basic Medical Sciences at Peking University have developed a targeted CD38 nanobody sequence using genetic engineering technology. They have optimized its structure, functionalized it with labeling, and conducted imaging and other evaluations, ultimately producing the CD38-targeted nuclear medicine small molecule diagnostic and therapeutic agent-68Ga-labeled nanobody NB381. The post-labeling quality control of the drug meets clinical trial requirements with a radiochemical purity (PCR) greater than 98% and in vitro stability not less than 90%.
  Preliminary PET imaging results of 68Ga-NB381 indicate that the nanobody is primarily concentrated in the kidneys, bladder, and MM.1S and Ramos or H929 tumors (CD38+). Additionally, the cold antibody NB381 significantly inhibits the uptake of 68Ga-NB381 in tumors, confirming the high specificity of this nanobody's binding to the CD38 protein.
  Other Names: 18F-FDG

SUMMARY:
Multiple myeloma (MM) predominantly affects the elderly, often presenting insidiously and with a rising incidence rate. Current diagnostic methods primarily rely on invasive bone marrow biopsies, which can lead to false-negative results if the biopsy site is improperly chosen. CD38 is significantly overexpressed on the surface of malignant plasma cells in MM, making it a characteristic tumor biomarker for this disease.

Addressing the limitations in specificity and sensitivity of traditional PET imaging agents, this project is dedicated to developing a new type of nanobody PET/CT imaging probe, 68Ga-NB381, which possesses high affinity and targets CD38. This probe, which is an intellectual property of our institution, aims to enhance the accuracy and specificity of early MM diagnosis. In terms of clinical evaluation, the project will implement a comprehensive assessment process including case selection, collection of baseline information, high-precision imaging, expert-level image interpretation, and follow-up studies, comparing directly with traditional 18F-FDG imaging to thoroughly verify the specificity and safety of 68Ga-NB381. This lays the groundwork for the clinical translation of this radiopharmaceutical in China. Furthermore, the project contributes to formulating more effective precision treatment plans based on CD38 expression levels and provides evidence for monitoring the therapeutic effects of daratumumab, a drug also targeting CD38. This makes the project of significant academic value and clinical importance, thus promoting the development of personalized treatment strategies.

DETAILED DESCRIPTION:
Multiple myeloma (MM) commonly occurs in the elderly and often remains undetected until it reaches an advanced stage. With the aging population in China, the incidence of MM is on the rise, now surpassing that of acute leukemia. Clinically, MM is characterized by bone destruction and lacks specificity; diagnosis primarily relies on bone marrow biopsies that detect an increase in clonal plasma cells, which are invasive and can yield false-negative results if the biopsy site is improperly selected. CD38 is significantly overexpressed on the surface of malignant plasma cells in MM, making it a characteristic tumor biomarker for MM.

As the incidence of malignant tumors in China continues to increase, so does the clinical demand for radiopharmaceuticals. Addressing the limitations in the targeting of 18F-FDG in PET imaging, the development of new targeted nuclear medicine molecular probes is of significant academic value and clinical importance, particularly in monitoring the therapeutic effects of the CD38-targeted nanobody NB381, which offers unique advantages. This project uses a nanobody with high affinity for CD38 as the targeting moiety for the radiopharmaceutical, exploring the diagnostic efficiency of 68Ga-NB381 in patients with MM exhibiting high CD38 expression. This not only provides a basis for the early diagnosis of MM but also allows for the formulation of effective precision treatment strategies based on the CD38 expression profile in MM patients.

68Ga-NB381, a new CD38-targeted molecular probe labeled with 68Ga, can be used for the diagnosis and research of various malignancies expressing high levels of CD38, including MM. The probe is conjugated with 68Ga3+ using TOHP as a bifunctional chelator, with a simple labeling process that does not require purification, offering high in-vivo stability and significant radioactive accumulation in tumor sites in mouse models, resulting in superior imaging outcomes. This project will complete the automation of the 68Ga-NB381 labeling process and conduct quality control studies on the resulting radiopharmaceutical injection solution, establishing quality standards for this new PET probe and laying the foundation for its clinical translation in China. The project aims to provide 68Ga-NB381 PET/CT imaging studies to support the early diagnosis of CD38 high-expression malignancies, the formulation of treatment plans, and the assessment of therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of multiple myeloma who are scheduled to undergo bone marrow aspiration or tissue biopsy within the next 3 months; aged between 18 and 90 years; participants must fully understand and voluntarily participate in this study, and sign an informed consent form; must be able to independently comply with the examination procedures.
* Confirmed symptomatic multiple myeloma patients; aged over 18 years; participants must fully understand and voluntarily participate in this study, and sign an informed consent form; must be able to independently comply with the examination procedures.

Exclusion Criteria:

* Pregnant women
* Individuals who cannot understand the examination process or are unable to cooperate.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Specificity and Binding Efficiency of 68Ga-NB381 in CD38 Positive Tumors | For a single patient, imaging and analysis will be conducted within 24 hours post-injection; follow-up assessments for stability and biodistribution will be conducted at 1 week post-injection.
  Evaluate the specificity and binding efficiency of 68Ga-labeled NB381 nanobody in targeting CD38 positive tumors using PET imaging. The measure involves comparing the uptake of 68Ga-NB381 in CD38 positive tumors to non-target areas and assessing the ability of cold antibody NB381 to inhibit this uptake, thus confirming the high specificity of the nanobody for CD38 protein.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Kang, MD, Study Director — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
All case data are anonymized before data analysis; all case files and imaging data are stored in a specialized database, which only the principal investigator is authorized to access and read; all researchers must not disclose any information about any patient.

REFERENCES:
- [Background] Bosseckert H. [The thrombolysis therapy, its application and dosage. II. Indications and practical application]. Z Arztl Fortbild (Jena). 1966 Jul 15;60(14):841-7. No abstract available. German. PMID 5994170
- [Background] Shephard GS, Thiel PG, Sydenham EW, Vleggaar R, Alberts JF. Determination of the mycotoxin fumonisin B1 and identification of its partially hydrolysed metabolites in the faeces of non-human primates. Food Chem Toxicol. 1994 Jan;32(1):23-9. doi: 10.1016/0278-6915(84)90032-2. PMID 8132161
- [Result] Korf J. Intracerebral trafficking of lactate in vivo during stress, exercise, electroconvulsive shock and ischemia as studied with microdialysis. Dev Neurosci. 1996;18(5-6):405-14. doi: 10.1159/000111434. PMID 8940612
- [Result] Zhang X, Hu W, Zhao G, Zhang Z, Zhang X, Gui Y, Zhang X, Wei H. A flow dialysis cell for on-line measurement of glucose in fermentation broth. Chin J Biotechnol. 1993;9(3):161-70. PMID 8049347